CLINICAL TRIAL: NCT00978562
Title: Imaging Vascular Properties of Pediatric Brain Tumors Using DSC-MRI With Ferumoxytol (Code 7228) and DCE-MRI With Gadolinium in a Single Imaging Session: An NCI Sponsored Exploratory Trial
Brief Title: DSC-MRI With Ferumoxytol and DCE-MRI With Gadolinium in Imaging Vascular Properties in Younger Patients With Brain Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00005405; NCI-2015-00227 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1562; 2864; SOL-09064-LX; 813; 5405 (Other: OHSU Knight Cancer Institute); R01CA137488 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Childhood Brain Neoplasm; Recurrent Childhood Brain Neoplasm
MeSH Terms: interventions — Ferrosoferric Oxide; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (DSC-MRI with ferumoxytol, DCE-MRI with gadolinium) (Experimental): Patients receive ferumoxytol and gadolinium IV and then undergo DSC-MRI and DCE-MRI. An optional MRI without injection of a contrast agent may be obtained after 20-24 hours at the discretion of the clinician. Patients may receive up to 3 more scans at least 3 weeks apart over up to 2 years.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol Non-Stoichiometric Magnetite; Drug: Gadolinium

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo DSC-MRI
  Other Names: Dynamic Susceptibility Contrast-Enhanced MRI
Drug: Ferumoxytol Non-Stoichiometric Magnetite — Given IV
  Other Names: Feraheme; Ferumoxytol
Drug: Gadolinium — Given IV
  Other Names: Gd

SUMMARY:
This clinical trial studies dynamic susceptibility-weighted contrast enhanced magnetic resonance imaging (DSC-MRI) after administration of ferumoxytol and dynamic contrast-enhanced MRI (DCE-MRI) after administration of a gadolinium-based contrast agent (GBCA) in viewing the vessels of the brain in younger patients with brain tumors. Ferumoxytol is an experimental form of very small iron particles that are taken by the blood stream to cells adjacent and inside the tumor. These iron particles may make it easier to see the areas of the brain that are affected by tumor. Ferumoxytol may work better than standard GBCA in viewing the vessels of the brain and brain tumor on MRI. Using ferumoxytol and GBCA in the same MRI session may provide more information about tumor blood supply and the extent of the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the vascular properties of pediatric brain tumors using ferumoxytol for DSC-MRI and GBCA for DCE-MRI in pediatric brain tumor (proven or presumptive) patients in a single MRI session.

II. To describe evolving imaging characteristics of tumor vasculature using DSC-MRI with ferumoxytol and DCE-MRI with GBCA in pediatric brain tumor patients.

SECONDARY OBJECTIVES:

I. Compare and evaluate magnetic resonance angiogram (MRA) with ferumoxytol between different time points.

II. To describe number and size of tumors imaged. III. To assess histology and electron microscopy (EM) on tissue samples. IV. To demonstrate differences in patients with prior therapy versus (vs.) no prior therapy (radiation and/or chemotherapy).

OUTLINE:

Patients receive ferumoxytol and gadolinium intravenously (IV) and then undergo DSC-MRI and DCE-MRI. An optional MRI without injection of a contrast agent may be obtained after 20-24 hours at the discretion of the clinician. Patients may receive up to 3 more scans at least 3 weeks apart over up to 2 years.

After completion of study treatment, patients are followed up at approximately 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have either radiological (presumptive) or established (proven) histological diagnosis of a brain tumor or lesion
* Previously untreated participants must have a measureable lesion on an imaging study
* Participants undergoing active treatment, or who have completed treatment, will have radiographic abnormalities that may or may not be recurrent tumor
* Those participants requiring surgical intervention for diagnostic and/or therapeutic purposes as necessary for their disease are eligible; the tissue may be assessed by histology and/or EM for iron particles; only clinically indicated biopsy and/or surgery will be done
* Participants may have had prior therapy for the primary brain tumor, including surgery, radiotherapy or chemotherapy
* After entry into the study, participants agree to be followed for up to 6 weeks after the final infusion of ferumoxytol
* All participants, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Baseline MRI studies for participants receiving ferumoxytol must be performed within 16 weeks of study entry
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study treatment and for the duration of study treatment; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Participants with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Participants with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations, are not eligible; participants with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion
* Participants who are pregnant, lactating, or who suspect they might be pregnant are not eligible
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than 2.5 x upper limits of normal
* Glomerular filtration rate (GFR) < 50
* Participants who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to GBCA
* Participants with known hepatic insufficiency or cirrhosis
* Human immunodeficiency virus (HIV)-positive participants on combination antiretroviral therapy are ineligible
* Participants that have a known or suspected iron overload (genetic hemochromatosis or history of multiple transfusions)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by participant before receiving study drug/imaging | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.64 (3.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Vascular Properties of Pediatric Brain Tumors Using Dynamic Susceptibility-weighted Contrast Enhanced MRI (DSC-MRI) After Administration of Ferumoxytol
Description: Signal intensity, relative cerebral blood volume (rCBV) was measured. Relative CBV measurements were calculated from regions of interest (ROI) that were placed in regions of highest perfusion seen on the rCBV color overlay parametric maps.The mean of 3 regions of contralateral white matter was used as the internal reference standard. The size of the ROIs was kept constant (radius 1.5 mm). Parametric color overlay maps were analyzed using ImageJ software (NIH, Bethesda, MD, USA).
Time Frame: Up to 2 years
Population: 7 participants had both appropriate ferumoxytol and gadolinium scans available for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: mL/g
Groups:
- Ferumoxytol DSC MRI: Subjects undergo MRI with ferumoxytol (study drug) and gadolinium (standard contrast agent) in the same imaging session. Ferumoxytol is given first and DSC images obtained, followed by gadolinium, and DCE images are obtained.
Arm/Group | Ferumoxytol DSC MRI
Number analyzed (Participants) | 7
mL/g | .93 (1.44)

2. Primary Outcome: Vascular Properties of Pediatric Brain Tumors Using Dynamic Contrast-enhanced MRI (DCE-MRI) After Administration of a Gadolinium-based Contrast Agent
Description: Volume transfer coefficient reflecting vascular permeability of pediatric brain tumors using Dynamic Contrast-enhanced MRI (DCE-MRI) was measured. Subjects undergo MRI with ferumoxytol (study drug) and gadolinium (standard contrast agent) in the same imaging session. Ferumoxytol is given first and DSC images obtained, followed by gadolinium, and DCE images are obtained.
Time Frame: up to 2 years
Population: 7 participants had both appropriate ferumoxytol and gadolinium scans available for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: min^-1
Groups:
- Gadolinium DCE: Subjects undergo MRI with ferumoxytol (study drug) and gadolinium (standard contrast agent) in the same imaging session. Ferumoxytol is given first and DSC images obtained, followed by gadolinium, and DCE images are obtained.
Arm/Group | Gadolinium DCE
Number analyzed (Participants) | 7
min^-1 | .25 (.23)

3. Secondary Outcome: Histology (Only in Patients for Whom a Biopsy or Surgery is Scheduled Outside of This Protocol)
Description: Appropriate descriptive statistics will be estimated. Results will be posted at overall completion.
Time Frame: Up to 2 years
Population: Due to low enrollment and staffing issues, data was not collected for this outcome.
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Enhancing Lesions
Description: Appropriate descriptive statistics will be estimated. Results will be posted at overall completion.
Time Frame: Up to 2 years
Population: Due to low enrollment and staffing issues, data was not collected for this outcome.
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 0

5. Secondary Outcome: Tumor Vascularity
Description: Appropriate descriptive statistics will be estimated. Results will be posted at overall completion.
Time Frame: Up to 2 years
Population: Due to low enrollment and staffing issues, data was not collected for this outcome.
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 0

6. Secondary Outcome: Ultrastructure (Only in Patients for Whom a Biopsy or Surgery is Scheduled Outside of This Protocol)
Description: Appropriate descriptive statistics will be estimated. Results will be posted at overall completion.
Time Frame: Up to 2 years
Population: Due to low enrollment and staffing issues, data was not collected for this outcome.
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 0

7. Secondary Outcome: Volume of Enhancing Lesions
Description: Appropriate descriptive statistics will be estimated. Results will be posted at overall completion.
Time Frame: Up to 2 years
Population: Due to low enrollment and staffing issues, data was not collected for this outcome.
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed up to 2 years
Description: All grades of adverse events were collected using Common Terminology Criteria for Adverse Events_v3.0 (CTCAE) (http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm)
Groups:
- Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium): Patients receive ferumoxytol and gadolinium IV and then undergo DSC-MRI and DCE-MRI. An optional MRI without injection of a contrast agent may be obtained after 20-24 hours at the discretion of the clinician. Patients may receive up to 3 more scans at least 3 weeks apart over up to 2 years.
  Dynamic Contrast-Enhanced Magnetic Resonance Imaging: Undergo DCE-MRI
  Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging: Undergo DSC-MRI Ferumoxytol Non-Stoichiometric Magnetite: Given IV
  Gadolinium: Given IV
Arm/Group | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium)
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium) (N=14)
Shunt malfunction and revision (Nervous system disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (DSC-MRI With Ferumoxytol, DCE-MRI With Gadolinium) (N=14)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diplopia (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
teleangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Body aches (General disorders) | 1 (1)
Shunt infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No